CLINICAL TRIAL: NCT05515276
Title: The COVID-19 Pandemic Process Increase Latex Glove Use and Latex Allergy Complaints in Hospital Nurses? Survey Study
Acronym: COVID19LATEX
Status: Completed | Type: Observational
Sponsor: Kilis 7 Aralik University (Other)
Responsible Party: Principal Investigator, İslam Elagöz, Principal Investigator, Kilis 7 Aralik University
Other Study IDs: Kilis 7 Aralık Üniversitesi
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: COVID-19 Pandemic; Nurse's Role; Allergy; Latex Allergy
Keywords: Latex Allergy; Latex Gloves; Corona virus disease; Nursing
MeSH Terms: conditions — COVID-19; Hypersensitivity; Latex Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Global guidelines recommend the use of personal protective equipment due to the high risk of contagiousness of COVID-19 disease. The increase in COVİD-19 patients in the last two years has increased the rate of use of latex gloves in nurses. It is not known how the increase in the use of latex gloves affects the complaints of latex allergy in nurses.

Aim: The aim of this study is to determine the rates of latex glove use and allergic complaints related to the use of latex gloves during the COVID-19 pandemic in hospital nurses.

DETAILED DESCRIPTION:
Background: Global guidelines recommend the use of personal protective equipment due to the high risk of contagiousness of COVID-19 disease. The increase in COVİD-19 patients in the last two years has increased the rate of use of latex gloves in nurses. It is not known how the increase in the use of latex gloves affects the complaints of latex allergy in nurses.

Aim: The aim of this study is to determine the rates of latex glove use and allergic complaints related to the use of latex gloves during the COVID-19 pandemic in hospital nurses.

Materials and Methods: Ethical and legal permissions were obtained before starting the research. Research; It was conducted in a descriptive and cross-sectional manner at Hatay Training and Research Hospital between May 15 and June 15, 2021. The sample of the study consisted of 448 nurses who volunteered to participate in the study. The data of the study were collected with data collection forms created by the researchers as a result of literature reviews. The data of the research were collected by the online questionnaire method. Analysis of the data was analyzed with appropriate statistical methods in SPSS 21.0 program. p<0.05 value was accepted for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Working as a nurse in Hatay Training and Research Hospital, Working in Hatay training and research hospital for the last month according to the date of the research
* Nurses who volunteered to participate in the study were included in the study.

Exclusion Criteria:

* Nurses who want to leave the study at any stage of the study after being included in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population of the study consisted of nurses working in Hatay Training and Research Hospital, and the sample consisted of nurses who met the inclusion criteria and volunteered to participate in the study. As a result of the research, 74.68% of the universe was reached. The sample size of the study was calculated in the G* Power 3.1.9.7 program, and a pyrori calculation was made according to the Mc Nemar test from the Exact test family. Cohen's d medium effect size was used in the calculation (Cohen J 1998). When the calculation is made such that odds ratio = 1.5, α error = 0.05, β error = 0.20, power = 0.80, effect size = 0.5 with the bidirectional hypothesis, the nurse to be sampled number was determined as N=398. The sample of the study (N=448) consisted of nurses.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Identifying Information Form: | 2023
  The identifying information form consists of questions aimed at determining the age, gender, education status, department of work, nursing experience, experience in the last working department, glove selection, family history of atopy, personal history of atopy, crossfood allergies, latex glove usage, duration of glove use in a day, number of invasive procedures, presence of diagnosed latex allergy, measures taken to prevent latex allergy, awareness of nonlatex gloves, and complaints after contact with latex-containing products.
Allergic Symptoms Evaluation Form: | 2023
  The form consists of questions aimed at determining skin reactions and allergic symptoms such as itching, redness, swelling, hives, lesions, rash, contact dermatitis, swelling 7 around the mouth and throat, nasal discharge, itching, sneezing, itching, redness, watering of the eyes, shortness of breath, coughing, wheezing, fainting, feeling of faintness, loss of consciousness, thinking that existing symptoms are related to work, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Islam, Kilis, Turkey (Türkiye)